CLINICAL TRIAL: NCT03324737
Title: Primary Prevention of Type 2 Diabetes: A Randomized Control Trial With Interactive Smartphone App to Restore Optimal Weight in Women With Recent Gestational Diabetes
Brief Title: Smartphone App to Restore Optimal Weight in Women With Recent Gestational Diabetes
Acronym: SPAROW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NMRC/HSRG/0071/2016
Record Dates: First submitted 2017-10-16; First posted 2017-10-30 (Actual); Last update posted 2019-08-08 (Actual); Status verified 2019-07

CONDITIONS: Gestational Diabetes; Weight Loss; Diet Habit
Keywords: Prevention; Smartphone application; Randomized control trial
MeSH Terms: conditions — Diabetes, Gestational; Weight Loss; Feeding Behavior

STUDY DESIGN:
Intervention Model Description: A prospective Randomized Control Trial will be conducted to compare an INTERACTIVE SMARTPHONE APP versus STANDARD care to optimize post-delivery weight in women with recent GDM. The aim is to reduce diabetes and cardiometabolic risk.
  During the antenatal period, subjects will be informed about the study during regular NUH nurse-led dietary counseling sessions. After delivery, women will be offered the opportunity to join the study. Informed consent will be obtained before discharge from hospital post-delivery. An appointment will be given for the first study visit at 6 weeks post-delivery.
Masking Description: The subjects who participate in the study may be seeing the doctors or allied health professionals involved in this study at the clinic. However, recruitment will not be done by them though they will help to improve the awareness of such a study to their patients. There will be no coercion involved as the subjects have the full autonomy to decide if they wish to participate.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Care Arm (No Intervention): Subjects in the standard care arm will be informed of their increased risk of developing type 2 diabetes in the future, and given general lifestyle verbal advice to maintain a healthy weight, eat a well-balanced diet and do regular exercise during their 6 week postnatal visit. Women found to have impaired fasting glucose (6.1-6.9 mmol/L) or impaired glucose tolerance (2H post glucose of 7.8-11.0 mmol/L) will be issued a letter reinforcing lifestyle changes namely weight loss (if raised BMI), diet, exercise, and encouragement to consult a family physician to discuss the appropriateness of starting medications that can prevent the progression to type 2 diabetes, or restore the blood glucose to normal levels. Those with a normal OGTT result will just be informed that it is normal.
- Interactive Smartphone App Arm (Active Comparator): Participants will download the INTERACTIVE SMARTPHONE APP and will be briefed on its use by our team of nutritionists/dieticians, exercise physiologists and life style coaches. Weight: Participants will be reminded that the goal is satisfactory weight loss.
  NUH occupational therapist-trained lifestyle coaches, exercise physiotherapists, and clinical nutritionist/ dietician will interact with participants through real-time chats channels via the APP; all culturally appropriate and customized to the Singapore context.
  Interventions: Device: Interactive Smartphone App

INTERVENTIONS:
Device: Interactive Smartphone App — There are six main components to the APP.
  * Goal Setting: personalizes diet, activity, and weight loss goals for patients based on their starting point.
  * Food choices and recommendations: App has an automated and immediate recommendation of foods if the choice selected from food database is not optimal. It has a calorie and nutrients tracker to enable patients to track their food intake.
  * Activity and steps tracker: App has a pedometer to count physical activity and steps to enable patients to track their progress towards goals.
  * Interactive video lessons: App has video lessons pushed weekly to the patient according to her needs. The videos encompass aspects of diet, lifestyle and behavior management.
  * Healthcare Professionals Support: App has a chat channel to enable interaction between participants and healthcare professionals.
  Arms: Interactive Smartphone App Arm

SUMMARY:
Gestational diabetes (GDM) complicates about 20% of pregnancies in Singapore. These women are at high risk of developing type 2 diabetes years after pregnancy; seven times more likely than normal. Achieving a healthy weight post-delivery is key to reduce the risk of future diabetes. This study, from a multidisciplinary team, intends to create a unique seamless care model to restore optimal weight post-delivery in women with recent GDM. The innovation examined in this randomized control trial is an INTERACTIVE SMARTPHONE APP. The APP monitors weight, dietary habits, and exercise activity patterns, gives feedback, and provides practical personalized lifestyle coaching that is culturally appropriate and customized to the Singapore context. If efficacy is confirmed in this RCT, the APP can be easily scaled up as a cost-effective way to potentially prevent or delay the onset of type 2 diabetes in Singaporean women. Additionally, measurement of markers of cardiometabolic risk will give indications on future cardiovascular health, utilizing an underused opportunity to improve women's health.

DETAILED DESCRIPTION:
About 20% of pregnant Singaporean women are diagnosed with gestational diabetes (GDM), defined as the onset of glucose intolerance that is first recognized in pregnancy. These women are at seven times higher risk of developing type 2 diabetes in the future. About 20 - 50% of women who were diagnosed with GDM during their pregnancies eventually develop type 2 diabetes, with resultant huge health care costs for Singapore and other countries globally. The Diabetes Prevention Program Study has shown that lifestyle changes resulting in modest weight loss are effective in preventing type 2 diabetes in women with a history of GDM. The investigators estimate that about 50% of all type 2 diabetes in women in Singapore occurs when they have a history of GDM and represent a sizeable subpopulation where primary prevention could have a highly significant national impact. Preliminary data indicates that after birth, women with GDM are overwhelmed with care for the newborn and tend to neglect their own health needs. They welcome reminders and coaching but are time-challenged and cannot attend regular on-site lifestyle coaching sessions.

Hypothesis:

1. Use of an INTERACTIVE SMARTPHONE APP that can track weight, diet and activity linked to an interactive lifestyle coaching intervention can restore optimal weight in women with recent GDM. The team hypothesizes that at 4 months post-delivery, participants in the intervention arm will have significantly higher probability of returning to weight at the start of pregnancy, a significantly improved cardiometabolic status and overall lower risk profile for type 2 diabetes development compared with those receiving standard care (control).
2. The use of this INTERACTIVE SMARTPHONE APP is cost-effective from the perspective of the Singapore healthcare system.

Aims:

1. To conduct a randomized control trial to examine the efficacy of an INTERACTIVE SMARTPHONE APP, customized for Singaporean women with recent GDM, in optimizing post-delivery weight and metabolic profiles compared with standard care.

   Primary outcome:
   * Restoration of booking weight if previous booking BMI ≤ 23
   * Weight loss of 5% with respect to booking weight if BMI > 23

   Secondary outcomes:

   - Improved cardiometabolic and inflammatory markers: fasting and 2h post-glucose load plasma glucose in an oral glucose tolerance test, HbA1C, advanced glycation end-products, C-peptide, HOMA-IR, lipid profile, liver function, hsCRP, IL-6.
2. Evaluate the relative cost-effectiveness of this INTERACTIVE SMARTPHONE APP compared to standard care within the Singapore healthcare system in terms of improvements in quality of life, feasibility, acceptability, scalability and sustainability.

ELIGIBILITY:
Inclusion Criteria:

* Female aged 21 years and above
* Plans to deliver in NUH
* Diagnosed with GDM antenatally (between 24-34 weeks gestation) defined using the 2013 World Health Organization criteria (fasting plasma glucose = 5.1 mmol/L, plasma glucose at 1H <10 or plasma glucose at 2H post 75gm glucose load of =8.5 mmol/L)
* Has a smartphone and able to independently use a smartphone app
* Willing to provide a blood sample
* Able to give written informed consent
* Able to speak and read English

Exclusion Criteria:

* Subjects with type 1 and/or type 2 diabetes (including suspected cases diagnosed by an abnormal oral glucose tolerance test in the 1st and early 2nd trimesters of pregnancy)
* drugs that affect glucose or lipid metabolism (e.g. systemic steroids, metformin, insulin, statins, orlistat)
* terminal or life threatening condition
* physical or mental condition that would prevent completion of a majority of study instruments.

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2017-11-16 (Actual); Primary Completion 2019-06-07 (Actual); Study Completion 2019-06-07 (Actual)

PRIMARY OUTCOMES:
Weight at 4 months post-delivery | 4 months
  Satisfactory weight is defined as return to weight at first booking visit (during 1st trimester) if booking BMI ≤23. If the booking weight is high (BMI>23), the goal would be return to weight that is 5% lower than booking weight.

SECONDARY OUTCOMES:
Markers predictive of future type 2 diabetes and cardiometabolic risk | 4 months
  Fasting and 2h post-glucose load plasma glucose in an oral glucose tolerance test, HbA1C, advanced glycation end-products, C-peptide, HOMA IR, lipid profile, liver function; and inflammatory risk: hsCRP, IL-6
Dietary assessment | 4 months
  Food Diary over 3 days to monitor the calorie intake and eating habits of the subject.
Subject's Self Efficacy to Regulate Exercise | 4 months
  The scale is devised by Bandura, and participants have to rate their degree of confidence in performing the described situations with a number from 0 to 100. The higher the value, the greater confidence the subject has in doing the activity.
Subject's Self Efficacy to Regulate Eating Habits | 4 months
  The scale is devised by Bandura, and participants have to rate their degree of confidence in performing the described situations with a number from 0 to 100. The higher the value, the greater confidence the subject has in doing the activity.
Subject's response to the research study using the Health Education Impact Questionnaire | 4 months
  A comparison between subjects' responses in the control and intervention arm, through a series of questions with 4 options - strongly disagree, disagree, agree, or strongly agree.
Subject's medical outcomes assessed through RAND-12 Item Health Survey | 4 months
  A comparison between subjects' responses in the control and intervention arm, through a series of questions about how she feels regarding aspects of her health and life. Questions are all multiple choice questions.
Subjects' health expenditure | 4 months
  A comparison between subjects' expenditure in the control and intervention arm, to find out the cost effectiveness of the study. Bill sizes and monetary expenditure (in dollars) will be calculated for every individual to find the amount she has spent on healthcare postnatally, due to GDM in her pregnancy.
DNA | 4 months
  DNA will be extracted and stored for future gene association studies with respect to type 2 diabetes susceptibility loci.
Breastfeeding Status | 4 months
  Patients will be categorised into fully, partial or no breastfeeding

CONTACTS AND LOCATIONS:
Overall Officials: Eu Leong Yong, Principal Investigator — National University Hospital, Singapore
Locations (1):
- National University Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lim K, Chan SY, Lim SL, Tai BC, Tsai C, Wong SR, Ang SM, Yew TW, Tai ES, Yong EL. A Smartphone App to Restore Optimal Weight (SPAROW) in Women With Recent Gestational Diabetes Mellitus: Randomized Controlled Trial. JMIR Mhealth Uhealth. 2021 Mar 16;9(3):e22147. doi: 10.2196/22147. PMID 33724204
- [Derived] Lim K, Chi C, Chan SY, Lim SL, Ang SM, Yoong JS, Tsai C, Wong SR, Yew TW, Tai ES, Yong EL. Smart Phone APP to Restore Optimal Weight (SPAROW): protocol for a randomised controlled trial for women with recent gestational diabetes. BMC Public Health. 2019 Oct 15;19(1):1287. doi: 10.1186/s12889-019-7691-3. PMID 31615456

DOCUMENTS (1):
  • Study Protocol (2017-11-01): https://cdn.clinicaltrials.gov/large-docs/37/NCT03324737/Prot_001.pdf